CLINICAL TRIAL: NCT05983315
Title: Prospective Assessment of CONECCT's Classification for Histological Predictive Diagnostic Value in Conducting Therapeutic Choice for Colorectal Lesions. Pro-CONECCT
Brief Title: Prospective Assessment of CONECCT's Classification for Colorectal Lesions.
Acronym: pro-CONECCT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0780
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
Keywords: diagnostic tool; colorectal cancer; therapeutic choice guidance; CONECCT
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CONECCT's classification assessment: Every patient who needs diagnostic colonoscopy because of digestive symptoms, medical or family history of colorectal cancer/polyps, positive colorectal screening test, acromegaly or referred by another gastroenterologist upon discovery of colorectal polyp after colonoscopy can join the cohort of this study and can get CONECCT's classification histological assessment of their neoplastic lesion by experienced endoscopist.

SUMMARY:
Colorectal neoplastic lesion endoscopic characterization is a key element for histological predictive diagnostic value in conducting best appropriate resection choice. Six classifications are necessary for fully correct characterization of different colorectal lesions. Nonetheless, it can be tricky to use so many diagnostic tools with so many subcategories in the 6 existing classifications. That's why we decided to integrate all 6 existing classification validated factors in one single chart (CONECCT chart) allowing to both predict histological diagnostic value and to propose the best appropriate resection strategy. A previous prospective and multicentre study with all French medical residents in gastroenterology was conducted in order to prove pedagogic interest of this diagnostic tool. Each student was asked to review 20 files with lesion pictures before and after lecture about CONECCT chart. This allowed us to prove that this diagnostic tool could significantly improve both histological predictive diagnostic value and therapeutic choice by French medical residents and gastroenterologists. Our hypothesis is that CONECCT's classification can improve predictive diagnostic value of colorectal lesions in over 80% of cases. Now that pedagogic interest of this diagnostic tool has been proven, we would like to carry out a larger prospective assessment in term of performance (value) of this instrument in order to both facilitate endoscopic characterization and allow a most appropriate diagnostic and therapeutic management of each colorectal lesion category.

ELIGIBILITY:
* Inclusion Criteria :

  * both gender patients even or older than 18 years old
  * patient in need of proven diagnostic or therapeutic colonoscopy for colorectal lesion resection
  * patient with French Health Insurance coverage
  * obtaining of oral non opposition to research after loyal, clear and complete delivery of information
* Exclusion Criteria :

  * previous attempt of lesion resection by mucosectomy
  * patient with a metastatic lesion diagnosed prior to colonoscopy
  * patient with no colorectal lesion
  * adenomatous or sessile serrated polyposis syndrome
  * patient with bowel chronic inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient who needs diagnostic colonoscopy because of digestive symptoms, medical or family history of colorectal cancer/polyps, positive colorectal screening test, acromegaly or referred by another gastroenterologist upon discovery of colorectal polyp after colonoscopy can join the cohort of this study.
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Correlation between endoscopic CONECCT's classification | Time point can be reached either 2 weeks after endoscopic resection at V1 or between 2-4 months later in case of surgery at V3
  assessed by one of research site operators and final histology reading of neoplastic lesion by anatomopathologist:
  * CONECCT 0E : neuroendocrine tumor
  * CONECCT IH : hyperplastic polyp
  * CONECCT IS : sessile serrated lesion with or without dysplasia
  * CONECCT IIA : low or high grade adenoma
  * CONECCT IIC : low or high grade adenoma or intramucosal or submucosal <1000 micron adenocarcinoma
  * CONECCT III : deep invasive submucosal > 1000 microns adenocarcinoma

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, France